CLINICAL TRIAL: NCT07150481
Title: Effect of Intravenous Lidocaine Infusion on Postoperative Inflammatory Response in Patients Undergoing Laparoscopic Cholecystectomy: A Randomized Double Blind Controlled Clinical Trial
Brief Title: Intraoperative Lidocaine Infusion
Acronym: IV
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Yahia Mohammd El-hagagy, Lecturer of anesthesia and intensive care, faculty of medicine, Assiut university., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Afaf Radi
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Enhanced Recovery After Anesthesia
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: group L: lidocaine IV infusion group C: normal saline 0.9% IV infusion
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group L (Active Comparator): IV Lidocaine infusion:
  Interventions: Drug: IV Lidocaine infusion
- Group C (Placebo Comparator): IV normal saline
  Interventions: Drug: IV normal saline

INTERVENTIONS:
Drug: IV Lidocaine infusion — 2 mg/kg/h (the total dose of lidocaine per hour will be calculated and add to normal saline 0.9% to total volume 50 ml and infused by a rate 50 ml/h till the end of the procedure
  Arms: Group L
Drug: IV normal saline — IV normal saline 0.9% , rate 50 ml/h
  Arms: Group C

SUMMARY:
This study aims to evaluate the analgesic and anti-inflammatory effect of perioperative intravenous lidocaine infusion and in turn the return of gastric motility in patients undergoing elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is considered a minimally invasive procedure; however, it still provokes a measurable systemic inflammatory response. This reaction is primarily driven by factors such as tissue manipulation, peritoneal insufflation, and surgical stress. C-reactive protein (CRP), a widely validated acute-phase reactant, serves as a reliable biomarker to monitor postoperative inflammation, typically peaking within 24 to 48 hours following surgery. Other inflammatory markers such as white blood cell (WBC) count, neutrophil-to-lymphocyte ratio (NLR), and interleukin-6 (IL-6) also exhibit perioperative changes, reflecting the underlying cytokine-mediated stress response. Monitoring these biomarkers provides insight into the extent of tissue injury and can help predict postoperative recovery or complications. Therefore, modulating the inflammatory response-such as through intravenous lidocaine infusion-may improve postoperative outcomes, including pain control, gastrointestinal recovery, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 - 60 years
2. Elective laparoscopic cholecystectomy for symptomatic cholelithiasis or chronic cholecystitis
3. ASA physical status I-II
4. BMI < 35 kg/m2
5. Preoperative CRP <20 mg/L
6. Informed consent provided

Exclusion Criteria:

1. Acute cholecystitis or biliary pancreatitis
2. Conversion to open surgery
3. Pre-op CRP >20 mg/L
4. Allergy to lidocaine or local anesthetics
5. Known hepatic or renal dysfunction
6. Chronic inflammatory conditions
7. Current immunosuppressive therapy
8. Cardiac arrhythmias or heart block without pacemaker
9. ASA physical status III, IV or above
10. Pregnancy or breastfeeding
11. Psychiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative CRP level | postoperative day 1 (24 hours postoperative)
  measurement of Postoperative CRP level

SECONDARY OUTCOMES:
Pain scores (VNS) | 2, 6, 12, 24 hours
  verbal numerical scale from 0-10. (0 = no pain, 10 = worst imaginable pain The patient verbally reports the number that best reflects their pain intensity.
GIT motility | within 24 hours
  Time to first pass of faeces or flatus/bowel movement
Postoperative complications | within 48 hours
  nausea, vomiting, ileus, infection
Time to ambulation | within 48 hours
  time of patient discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Noha Y Mohamed, MD, Principal Investigator — Lecturer in anesthesia and intensive care department, faculty of medicine,; Noha Y Mohammed, MD, Principal Investigator — Lecturer in anesthesia and intensive care department, faculty of medicine,
Locations (1):
- Assiut university main hospital, Asyut, Assiut Governorate, Egypt,, Egypt

IPD SHARING:
Plan to Share IPD: No